CLINICAL TRIAL: NCT04579081
Title: Post Market Clinical Follow-up (PMCF)Study of the Contour Neurovascular SystemTM
Status: Withdrawn | Type: Observational
Why Stopped: This study has not been started. The Sponsor has decided not to pursue this study.
Sponsor: Cerus Endovascular, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DNX090-03
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Contour Neurovascular System — Intrasaccular flow disruptor/divertor

SUMMARY:
Cerus Endovascular is sponsoring a prospective, multi-center PMCF to document the safety and performance of the Contour Neurovascular System™ (hereinafter "Contour") in normal medical use.

DETAILED DESCRIPTION:
The primary objective of this study is to document the safety and performance of the "Contour Neurovascular System™. The data from the study will be reported as a Post Market study to the Notified Body as part of the Post Market Surveillance (PMS) and Post Market Clinical Follow-up (PMCF) plan.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient indicated for treatment of a single, unruptured aneurysm is according to the national/international guidelines.

  2. Age 18 years or older at screening. 3. Patient suitable for non-emergency endovascular embolization of saccular IAs.

  4. IA located at a bifurcation in the anterior or posterior circulation with dimensions consistent with implant size selection guidelines included in the IFU for Contour.

  5. Patient has the necessary mental capacity to participate and is willing and able to participate in the study for the duration of the study follow-up and is able to comply with study requirements.

  6. Patient is able to give their informed consent. This must be demonstrated by means of a personally signed and dated informed consent document indicating that the subject has been informed of and understood all pertinent aspects of the study.
* Exclusion Criteria

  1. Ruptured aneurysm.
  2. Patient anatomy or physiology considered unsuitable for endovascular treatment.
  3. Contraindication for arterial access.
  4. Largest measured IA equatorial diameter >8.5 mm or <2 mm.
  5. Largest measured IA neck diameter >8 mm or <2 mm.
  6. Target IA contains other devices/implants that could interfere with proper placement of the Contour device (e.g., coils).
  7. Known allergy to platinum, nickel or titanium.
  8. Known allergy or intolerance to contrast agents.
  9. Contraindication to anticoagulants or platelet inhibitor medication.
  10. In the opinion of the investigator, any other medical issue within the brain that precludes the device implantation such as brain surgery, radiation in the target area of intervention, acute traumatic craniocerebral injury, etc.
  11. Other medical conditions that cause an inability to comply with study requirements and/or that could increase the risk of neurovascular procedures or death within 2 years (e.g., liver failure, cancer, heart failure, chronic obstructive pulmonary disease, immunosuppression, neural disease, substance abuse and hematologic disorders etc.).
  12. Participating in another study with investigational devices or drugs that would confound the effects of the study outcomes.
  13. The presence of a condition that may create unacceptable risk during the aneurysm embolization procedure.
  14. Female patient who is pregnant or breastfeeding.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with enraptured bifurcated intracranial aneurysms.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with non-accidental death cause or any major ipsilateral stroke within the first 30 days after treatment or major ipsilateral stroke or death due to neurological cause from day 31 to final follow-up visit per standard of care). | 1 year
  Primary Safety Endpoint
Aneurysm occlusion rate on the follow-up angiogram as reported by the investigator." "Success will be defined as complete occlusion demonstrated by a Grade 1 using the Raymond Roy (RR) Scale. | 1 year
  Primary Performance Endpoint

IPD SHARING:
Plan to Share IPD: No